CLINICAL TRIAL: NCT06422000
Title: Pentoxifylline Versus Probiotic as Adjuvant Therapy for Preterm Neonates With Necrotizing Enterocolitis
Brief Title: Effect of Pentoxifylline Versus Probiotic on Preterm Neonates With Necrotizing Enterocolitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Alaa Mohamed Ahmed Rowisha, clinical pharmacist, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pentoxifylline probiotic NEC
Record Dates: First submitted 2022-11-11; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Necrotizing Enterocolitis
MeSH Terms: conditions — Enterocolitis, Necrotizing | interventions — Pentoxifylline

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (group I) (No Intervention): will include 25 preterm neonates with NEC who will receive traditional therapy of NEC including antibiotics and normal incubator care measures
- pentoxifylline group (group II) (Active Comparator): will include 25 preterm neonates with NEC who will receive traditional therapy of NEC in association with IV pentoxifylline at a dose of 30 mg/kg given over 6 hours daily (Schüller et al., 2020) until discharge from the unit after clinical and laboratory improvement .
  Interventions: Drug: Pentoxifylline
- probiotic group (group III) (Active Comparator): will include 25 preterm neonates with NEC who will receive traditional therapy of NEC in association with probiotics sachets supplementation, in the form of lyophilized lactic acid bacteria each Aluminium stick pack contains 100 mg ( Meyer et al., 2020) Probio Tec BB12-Blend 30- IF* (SANDOZ®.) mixed with 10 ml sterile water and given by Ryle tube once daily until discharge from the unit after clinical and laboratory improvement .
  Interventions: Drug: Probiotic Formula

INTERVENTIONS:
Drug: Pentoxifylline — Pentoxifylline 30 mg/kg given over 6 hours daily
  Other Names: group 2 (Pentoxifylline group)
  Arms: pentoxifylline group (group II)
Drug: Probiotic Formula — probiotics sachets supplementation, in the form of lyophilized lactic acid bacteria each Aluminium stick pack contains 100 mg ( Meyer et al., 2020) Probio Tec BB12-Blend 30- IF* (SANDOZ®.) mixed with 10 ml sterile water and given by Ryle tube once daily until discharge from the unit after clinical and laboratory improvement .
  Other Names: group 3 (Probiotic group)
  Arms: probiotic group (group III)

SUMMARY:
The aim of this study is to evaluate the effectiveness of pentoxifylline versus probiotics supplementation as adjuvant therapy for preterm neonates with necrotizing enterocolitis.

DETAILED DESCRIPTION:
This randomized clinical trial includes 75 preterm infants who met the inclusion criteria for stage I and stage II NEC. Patients are allocated randomly into three groups (each included 25 neonates); group I (traditional therapy group) received antibiotics according to culture and sensitivity results, group II (pentoxifylline group) received antibiotics and IV pentoxifylline at a dose of 30 mg/ Kg given over 6 hours daily until discharge from the unit, and group III (probiotics group) received antibiotics and probiotics sachets supplementation in a dose of 100 mg mixed with 10 ml sterile water and given by Ryle tube once daily until discharge. The serum level of high-mobility group box protein 1 (HMGB-1), intestinal fatty acid binding proteins (I-FABP), and total antioxidant capacity (TAC) were measured on admission and at discharge.

ELIGIBILITY:
Inclusion Criteria:

* Male and female preterm neonates less than 37 weeks gestational age
* Suffering from necrotizing enterocolitis (NEC), according to Modified Bell's system which was first proposed by Bell et al., 1978 as stage I (suspected), II (proven) .
* Diagnosis of NEC depends on; history, physical examination, laboratory and radiographic findings .
* Signs and symptoms of NEC (at least three or more ), including; unstable temperature, apnea, increased residual milk in stomach, mid abdominal distension, vomiting coffee-like substances, bloody stool
* Laboratory findings including; thrombocytopenia, hypernatremia, metabolic acidosis, neutropenia and leukocytosis.
* Anterior posterior abdominal radiograph is used for diagnosis in which pneomatosis intestinalis in stage II NEC

Exclusion Criteria:

* Term and post term neonates
* Neonates with congenital infections
* Neonates with major congenital anomalies
* Neonates with stage III NEC

Max Age: 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Mortality rate | 2 months
  record mortality rate in each group during treatment
complications and side effects | 2 months
  record any complications or side effects of the treating drugs
Inflammatory parameter | 2 months
  Change in serum C-reactive protein at baseline and after 2 months

SECONDARY OUTCOMES:
change in serum high-mobility group box protein 1 (HMGB1) | 2 months
  blood sample will be collected at baseline and after 2 months
change in serum Intestinal fatty acid binding protein (I-FABP). | 2 months
  blood sample will be collected at baseline and after 2 months
change in serum total antioxidant capacity (TAC) | 2 months
  Blood sample will be collected at baseline and after 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Sahar Hegazy, MD, Study Director — professor and head of clinical pharmacy department, faculty of Pharmact, Tanta University, Egypt
Locations (1):
- Tanta University, Tanta, El Gharbia, Egypt